CLINICAL TRIAL: NCT07072494
Title: Clinical Study on the Efficacy and Safety of CD19 CAR-T Cell Infusion as Consolidation Therapy in Adolescent and Adult Patients With Acute B-Lymphoblastic Leukemia Who Are Ineligible for Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: CD19 CAR-T Cell Infusion as Consolidation Therapy in Adolescent and Adult Patients With Acute B-ALL Ineligible for Allogeneic HSCT: A Clinical Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-394-01
Record Dates: First submitted 2025-03-24; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Chimeric Antigen Receptor T-Cell Immunotherapy; CD19; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Consolidation therapy with CAR-T cells was performed after induced remission (Experimental): For autologous intravenous infusion only, the recommended dose is 0.5×108 CAR-T live cells, and the dose range is 0.25~0.5×108 CAR-T live cells (±20%, i.e. 0.2-0.6×108 CAR-T live cells)
  Interventions: Drug: CD19 CAR-T cells injection

INTERVENTIONS:
Drug: CD19 CAR-T cells injection — Lymphodepleting pre-treatment will begin one week before the CAR-T cell infusion to reduce the burden of abnormal immune cells in the body, creating a favorable environment for the infused CAR-T cells. The suggested pre-treatment regimen is based on the FC regimen (Fludarabine + Cyclophosphamide).After the pre-treatment, patients will undergo CAR-T cell infusion, where the genetically modified T-cells are infused back into the patient's body.

SUMMARY:
This clinical study investigates a novel treatment option for adolescents and adults with acute B-lymphoblastic leukemia (B-ALL). While allogeneic hematopoietic stem cell transplantation (HSCT) is a standard therapy for leukemia, some patients are ineligible due to factors such as age, underlying medical conditions, or the absence of a suitable donor. For these individuals, CD19 CAR-T cell therapy is being evaluated as a potential consolidation therapy.

DETAILED DESCRIPTION:
This is an open-label, single-arm, prospective clinical study designed to evaluate the clinical effectiveness and safety of CD19-directed chimeric antigen receptor T (CAR-T) cell therapy as a consolidation treatment in adolescent and adult patients with acute B-ALL who are ineligible for allogeneic HSCT. The study is planned to be conducted over a period of three years, enrolling a total of 30 participants.The primary objective of this study is to assess the clinical effectiveness of CD19 CAR-T cell therapy as a consolidation therapy in achieving remission and improving survival outcomes in the specified patient population. Specifically, the study aims to:

Evaluate the efficacy of CD19 CAR-T cell therapy in achieving complete remission (CR) or minimal residual disease-negative (MRD-) status in patients with B-ALL.

Assess the safety and tolerability of the treatment, with a focus on key adverse events.

Eligible participants will receive CD19 CAR-T cell infusion following a standard lymphodepleting chemotherapy regimen. After infusion, patients will be closely monitored for both short-term and long-term outcomes. Safety Considerations:

Patients will be closely monitored for treatment-related toxicities. Early intervention strategies for CRS and neurotoxicity will be implemented as per established management guidelines. Supportive care, including corticosteroids and anti-cytokine therapies, will be available for severe toxicities.

This study seeks to provide valuable clinical evidence regarding the use of CD19 CAR-T cell therapy as a consolidation strategy for B-ALL patients who are not candidates for HSCT. By evaluating both efficacy and safety parameters, the study aims to contribute to the growing body of knowledge surrounding CAR-T therapies in hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has voluntarily agreed to participate, signed the informed consent form, and is willing and able to comply with scheduled visits, study treatment, laboratory tests, and other study procedures.
2. The subject has been clinically diagnosed with newly diagnosed or refractory/relapsed B-cell acute lymphoblastic leukemia (B-ALL), including Burkitt lymphoma leukemia and blast-phase chronic myeloid leukemia, and has achieved complete remission (defined as <5% bone marrow blasts, no peripheral blood blasts, and no extramedullary leukemia) after chemotherapy or immunotherapy, but is either ineligible for allogeneic hematopoietic stem cell transplantation (allo-HSCT), lacks a suitable donor, or declines transplantation.
3. Aged between 14 and 80 years (inclusive), male or female.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. At the time of screening, leukemia cells in the bone marrow or peripheral blood must be confirmed as CD19-positive by flow cytometry at initial or relapse diagnosis.
6. An expected survival of more than three months from the date of signing the informed consent form.
7. Satisfactory liver, kidney, cardiac, and pulmonary function, defined as:

   1. Creatinine ≤2× upper limit of normal (ULN);
   2. Left ventricular ejection fraction (LVEF) ≥50%;
   3. Blood oxygen saturation >92%;
   4. Total bilirubin ≤2× ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3× ULN.
8. Adequate venous access for cell collection and meeting the following hematologic criteria:

   Hemoglobin ≥80 g/L Absolute neutrophil count (ANC) ≥1.0 × 10⁹/L Platelet count ≥75 × 10⁹/L If the above criteria are not met, the investigator may determine eligibility for mononuclear cell collection.
9. Female subjects of childbearing potential must have a negative serum pregnancy test (women who have undergone surgical sterilization or have been postmenopausal for at least two years are considered non-fertile). Male and female subjects of reproductive potential must agree to use contraception during the study.

Exclusion Criteria:

1. Presence of mixed-lineage leukemia or biphenotypic leukemia.
2. Prior treatment with CAR-T cell therapy before screening or conditioning.
3. Patients with bone marrow failure syndromes associated with genetic disorders, such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndromes.
4. Any of the following viral infections:

   Hepatitis B virus (HBV) DNA detectable above the lower limit of quantification. Positive hepatitis C virus antibody (HCV-Ab). Epstein-Barr virus (EBV) or cytomegalovirus (CMV) DNA detectable above the lower limit of quantification.

   Positive human immunodeficiency virus (HIV) antibody test.
5. History of or current malignancy within the past five years (excluding patients with a low risk of recurrence after curative treatment and more than five years of follow-up, as determined by the investigator).
6. Any of the following cardiac conditions:

   New York Heart Association (NYHA) Class III or IV congestive heart failure. Severe arrhythmia requiring treatment or clinically significant conduction abnormalities on ECG, including QTc interval ≥480 ms (QTcB = QT/√RR).

   Uncontrolled hypertension despite standard treatment (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg) or pulmonary hypertension.

   Unstable angina. Myocardial infarction, coronary artery bypass grafting, or stent placement within six months before cell infusion.

   Clinically significant valvular heart disease. Other cardiac diseases deemed inappropriate for study participation by the investigator.
7. Uncontrolled epilepsy, a history of cerebrovascular ischemia/hemorrhage, cerebellar disease, or other active central nervous system (CNS) disorders.
8. Clinically significant pericardial or pleural effusion at screening.
9. History of deep vein thrombosis or pulmonary embolism within six months before screening.
10. Known hypersensitivity to any component of the study treatment.
11. Live vaccine administration within six weeks before screening.
12. Severe, uncontrolled, active infection at screening.
13. Participation in other interventional clinical trials and receipt of an investigational agent, including:

    An unapproved investigational drug within three months before cell infusion. A marketed drug within fewer than five half-lives before cell infusion.
14. Any other conditions deemed unsuitable for study participation by the investigator.
15. Physical or cognitive conditions that impair the ability to provide informed consent or comply with study procedures, or unwillingness or inability to adhere to study requirements.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-19 (Estimated); Primary Completion 2027-03-19 (Estimated); Study Completion 2027-08-19 (Estimated)

PRIMARY OUTCOMES:
Leukemia-Free Survival(LFS) | From Chimeric Antigen Receptor T-Cell infusion to relapse or death, assessed up to 12 months
  Relapse defined by ≥ BM blasts(ELN 2022)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol